CLINICAL TRIAL: NCT04832711
Title: A Community Study of the Risk for Obstructive Sleep Apnea and Respiratory Inflammation in an Adult Chinese Population
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jing MA, Prof.&MD, Peking University First Hospital
Other Study IDs: 2021-116
Record Dates: First submitted 2021-03-28; First posted 2021-04-06 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea; Inflammation; Exhaled Breath Condensate; Surveys and Questionnaires
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — exhaled breath condensate; plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the low-risk group for OSA: A Chinese translation of the BQ was used to classify subjects into high risk and low risk for OSA.
- the high-risk group for OSA: A Chinese translation of the BQ was used to classify subjects into high risk and low risk for OSA.

SUMMARY:
We aimed to investigate the relationship between obstructive sleep apnea (OSA) risk and respiratory inflammation evaluated by the exhaled breath condensate （EBC）interleukin-6 IL-6 and plasma SP-D, based on the Berlin questionnaire (BQ) screening values in an adult, urban community in Beijing, China.

Volunteers aged >40 years were recruited from the Shichahai community of central Beijing. Their general information and disease history were recorded. OSA risk was assessed using the BQ. IL-6 in EBC and plasma SP-D were detected by enzyme-linked immunoassay (ELISA)through specimens collected on fasting. The differences in IL-6 and SP-D contents between high-risk and low-risk groups for OSA were compared, and the factors affecting their contents were analyzed.

DETAILED DESCRIPTION:
Subjects

The volunteers were recruited residents from the Shi Cha Hai community of Beijing, China. The inclusion criteria included individuals aged ≥40 years who had stayed in the community for at least 3 years and who had provided informed consent.

In contrast, the exclusion criteria were patients with known severe diseases who could not cooperate with the study, such as severe psychiatric diseases, chronic liver disease, heart failure, autoimmune disease, and chronic kidney disease; a history of pulmonary lobectomy or lung transplantation; and drug abuse or alcohol addiction.

Questionnaire survey and physical examination Community volunteers were surveyed for general information (name, sex, age, height, weight, etc.), history of previous common diseases, medication use, history of smoking, history of alcohol consumption, and occupation. All surveys were filled in the case report form of the study. A Chinese translation of the BQ was used to classify participants as high risk and low risk for OSA. COPD were diagnosed by a portable spirometer (Vitalograph copd-6). Other investigated diseases were self-reported by participants based on previous diagnosis. Physical examination included blood pressure, height, and weight measurements.

Sample collection and storage Venous blood and EBC were collected between 9 AM and 12 AM after fasting for >10 hours. The plasma collected in EDTA anticoagulated blood collection tubes was separated by centrifugation at 2,000 g for 15 min and stored at -80℃. The EBC collection was performed using an EBC collector (model number, EBC-5; patent number, ZL 2019 2 1297152.7, China).

The EBC collection was conducted as follows: After resting for 15 minutes and cleaning the oral cavity with water, participants were instructed to wear a nose clip and breathe calmly through a mouthpiece with a one-way valve, which was connected to an electrical condenser. Participants were asked to breathe through the device for 15 minutes to obtain between 0.5 and 1.5 ml of condensate. After being pre-processed with argon flow of 0.25 L/min for 10 minutes, the condensate was immediately fractional packed and transferred to special tubes and stored at -80℃. EBC equipment, collection procedures, and preservation complied with European Respiratory Society standards on breath analyses .

Measurement of biomarkers Enzyme-linked immunosorbent assay (ELISA) kits were used to measure the biomarkers in both EBC and plasma.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included individuals aged ≥40 years who had stayed in the community for at least 3 years and who had provided informed consent.

Exclusion Criteria:

* the exclusion criteria were patients with known severe diseases who could not cooperate in the study, such as severe psychiatric diseases, chronic liver disease, heart failure, autoimmune disease, and chronic kidney disease, and a history of pulmonary lobectomy or lung transplantation and drug abuse or alcohol addiction.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The volunteers were recruited residents from the Shi Cha Hai community of Beijing, China.
Sampling Method: Non-Probability Sample
Enrollment: 1270 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Correlation between risk for OSA and inflammation | through study completion, an average of 3 year
  The levels of EBC IL-6 and plasma SP-D were detected by ELISA. The levels of EBC IL-6 and plasma SP-D between the high- and low-OSA risk groups were compared.

SECONDARY OUTCOMES:
Comorbidities, inflammation and risk of sleep apnea | through study completion, an average of 3 year
  The prevalence of hypertension, coronary heart disease, and diabetes in the high-risk group for OSA than in the low-risk group were explored.

CONTACTS AND LOCATIONS:
Locations (1):
- Jing Ma, Pro., Beijing, China

IPD SHARING:
Plan to Share IPD: No